CLINICAL TRIAL: NCT07334730
Title: A Prospective Analysis of the Effects of Holmium Laser Enucleation (HoLEP) and Thulium Laser Enucleation (ThuLEP) on Continence, Urethral Stricture, and Sexual Function in Benign Prostatic Hyperplasia
Brief Title: The Effects of Holmium Laser Enucleation and Thulium Laser Enucleation on Continence, Urethral Stricture, and Sexual Function in Benign Prostatic Hyperplasia
Acronym: EHTCUS
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Halil Tosun, Halil Tosun Assistant Proffessor, TC Erciyes University
Other Study IDs: COMP_AFTER_HOLEP_THULEP_26
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostate Obstruction (BPO)
Keywords: HOLEP; THULEP; BPO; Urinary Incontinence; Sexual Function; Urethral Stricture; Benign Prostate Obstruction; Benign Prostate Hyperplasia; Holmium; Thulium
MeSH Terms: conditions — Urinary Incontinence; Urethral Stricture; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Benign Prostatic Obstruction Patient Group: The effects of Holmium Laser Enucleation (HoLEP) and Thulium Laser Enucleation (ThuLEP) surgeries on continence, urethral stricture, and sexual function in patients with benign prostatic hyperplasia were investigated prospectively.

SUMMARY:
This study aims to evaluate the effects of Holmium Laser Enucleation of the Prostate (HoLEP) and Thulium Laser Enucleation of the Prostate (ThuLEP), performed for the treatment of benign prostatic hyperplasia (BPH), on the following parameters: urinary continence, development of urethral or bladder neck stricture, and sexual function, including erectile function, ejaculation, and libido.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a progressive condition commonly affecting men, characterized by lower urinary tract symptoms (LUTS) that increase in prevalence and severity with age. Although medical therapy is effective for many patients, approximately 5% experience symptom progression requiring surgical intervention. While transurethral resection of the prostate (TURP) has long been considered the standard surgical treatment, technological advancements have enabled the widespread use of anatomical endoscopic enucleation of the prostate (AEEP) employing various laser modalities. Among these, Holmium laser enucleation of the prostate (HoLEP) and thulium laser enucleation of the prostate (ThuLEP) are established minimally invasive techniques used in the surgical management of BPH.

Detailed Description

Recent studies have demonstrated comparable perioperative and functional outcomes between HoLEP and ThuLEP, with no significant differences reported in terms of urinary retention, stress urinary incontinence, bladder neck contracture, or urethral stricture formation. However, postoperative evolution of urinary continence, overactive bladder symptoms, and sexual function remains a clinically relevant concern, particularly regarding patients' quality of life. Despite the increasing use of laser-based enucleation techniques, comparative data focusing on continence status, urethral or bladder neck stricture development, and sexual function outcomes remain limited.

To reduce postoperative complications, several surgical technique modifications have been introduced, including en bloc enucleation, two-lobe and three-lobe techniques, as well as urethral mucosa-preserving approaches such as single-N and double-N techniques. These modifications aim to preserve periurethral and paracollicular tissues, particularly in proximity to the verumontanum, thereby potentially improving functional outcomes.

The prevalence of BPH continues to rise in the aging population, often accompanied by systemic comorbidities and the use of anticoagulant or antithrombotic medications, which are associated with an increased risk of postoperative bleeding and hemorrhagic complications. Consequently, there is a growing need to evaluate the long-term outcomes of minimally invasive surgical techniques in this patient population.

This study aims to address existing gaps in the literature by providing comparative data on the long-term functional outcomes of minimally invasive surgical approaches for BPH, thereby contributing to improved patient selection, surgical technique optimization, and postoperative quality-of-life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of benign prostatic hyperplasia (BPH).
* Indication for surgical treatment of BPH.
* Male patients aged 40-90 years.

Exclusion Criteria:

* Patients with active urinary tract infection (UTI).
* Patients at high risk who cannot undergo spinal or general anesthesia.
* Patients with uncontrolled bleeding diathesis.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Benign prostatic obstruction is a male-specific condition
Study Population: Adult male patients treated surgically for benign prostatic obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Postoperative Urethral Stricture or Urinary Incontinance | Within 6 months after surgery
  Postoperative urethral stricture was defined as a maximum urinary flow rate (Qmax) of less than 15 mL/s on uroflowmetry at the first postoperative month, accompanied by a voiding curve pattern consistent with urethral obstruction. Postoperative urinary incontinence was defined as the presence of patient-reported urge or stress-type incontinence at the first postoperative month, supported by an increased score on the International Consultation on Incontinence Questionnaire (ICIQ)

SECONDARY OUTCOMES:
Number of participants assessed for sexual function | within 6 months after surgery
  Patients' sexual function will be evaluated using the Male Sexual Health Questionnaire (MSHQ) and the International Index of Erectile Function-5 (IIEF-5) for both HoLEP and ThuLEP procedures.
Number of participants with surgery-related complications | Within 6 months after surgery
  Surgical technique-related complications were defined as intraoperative or early postoperative events, including postoperative bleeding, prostatic capsular injury, and bladder perforation, and were classified according to the Clavien-Dindo classification system.
Number of participants presenting with lower urinary tract symptoms | Within 6 months after surgery
  Lower urinary tract symptoms (LUTS) were categorized as storage and voiding symptoms. Storage symptoms included dysuria, nocturia, pollakiuria, and urge urinary incontinence, whereas voiding symptoms comprised weak urinary stream and delayed initiation of micturition. LUTS were assessed using the International Prostate Symptom Score (IPSS) and the International Consultation on Incontinence Questionnaire-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS).

CONTACTS AND LOCATIONS:
Overall Officials: HALİL TOSUN, Assistant Professor, Principal Investigator — TC Erciyes University; EMRE C. AKINSAL, Assoc. Prof., Study Chair — TC Erciyes University
Locations (1):
- Erciyes University Faculty of Medicine, Department of Urology, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No